CLINICAL TRIAL: NCT04353752
Title: The Natural History of Cystic Fibrosis in the Era of Next Gen Combination Modulator Agents: Novel Treatment Targets in an Evolving Disease
Brief Title: Observational Trial of the Longitudinal Effects of CFTR Modulator Drugs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Jewish Health (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: SAAVED19AO-PG
Record Dates: First submitted 2020-03-20; First posted 2020-04-20 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
CF patients enrolled in this protocol will be recruited from patients followed by the Adult CF Program at National Jewish Health. Patients will be selected based on planned use of a CFTR modulator by their primary physician. No patient will be started on (or will switch) CFTR modulator agents for the purpose of the study. After enrollment, biological samples may be collected at two different time points prior to treatment initiation. One set of samples will be collected at baseline health prior to CFTR modulator initiation or change. A second set of samples will be obtained in subjects at the time of acute pulmonary exacerbation, if one occurs prior to CFTR modulator initiation or change. Post CFTR modulator initiation study assessments will be obtained at least one month after starting treatment and continue up to 2 times a year (including during pulmonary exacerbations), in order to document longitudinal effects of therapies and changes in inflammatory biology over time. At the time of each biological sampling, blood, sputum sample, urine, and a quality of life assessment will be acquired in all enrolled subjects. In addition to demographic data, clinical data, such as quantitative microbiology and simple spirometry will be recorded at the time of sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CF with an eligible mutation for modulator treatment.
* Age 18 years old or older.
* Patient is starting a CFTR modulator as part of their clinical care or switching CFTR modulator therapy agents, pending FDA approval.
* Ability to perform reproducible Pulmonary Function Tests.
* Willingness to comply with study procedure and willingness to provide written consent.

Exclusion Criteria:

• Presence of a condition or abnormality that, in the opinion of the Principal Investigator (PI), would compromise the safety of the patient or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in this protocol will be recruited from patients followed by the Adult CF Program at National Jewish Health. The investigators project enrolling 80 subjects with diagnosed CF, 18 years of age or older, with eligible mutations for CFTR modulator therapies. Concomitant use of systemic steroids will be allowed, and typical co-infections or co-morbidities will not result in exclusion.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood inflammatory markers | Before initiation/change of CFTR modulator and after, on average 6 months apart
  Changes in host inflammation as measured in peripheral blood memory T cells
Change in sputum microbiology | Before initiation/change of CFTR modulator and after, on average 6 months apart
  Changes in the bacterial burden in sputum as measured by bacterial RNA

SECONDARY OUTCOMES:
Changes in lung function | Before initiation/change of CFTR modulator and after, on average 6 months apart
  Changes in lung function as measured by FEV1, % predicted
Changes in urine inflammatory marker | Before initiation/change of CFTR modulator and after, on average 6 months apart
  Changes in host inflammation as measured by urinary neutrophil gelatinase-associated lipocalin (NGAL)
Changes in quality of life | Before initiation/change of CFTR modulator and after, on average 6 months apart
  Changes in quality of life as measured by Cystic Fibrosis Questionnaire - Revised (CFQ-R)
Changes in hospitalizations | Before initiation/change of CFTR modulator and after, on average 6 months apart
  Changes in frequency/number of hospitalizations for treatment of pulmonary exacerbation

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No